CLINICAL TRIAL: NCT06416358
Title: A Phase IIa, Multi-center, Single-Arm, Open-Label Study to Evaluate the Efficacy of ALMB-0168 in Solid Tumor Patients With Bone Metastatic Whose Prior Standard Treatment Have Failed
Brief Title: A Study to Evaluate the Efficacy of ALMB-0168 in Solid Tumor Patients With Bone Metastatic Whose Prior Standard Treatment Have Failed
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: AlaMab Therapeutics (Shanghai) Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ALMB-0168-002
Record Dates: First submitted 2024-05-10; First posted 2024-05-16 (Actual); Last update posted 2024-05-16 (Actual); Status verified 2024-05

CONDITIONS: Advanced Solid Tumors With Bone Only Metastasis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- ALMB-0168 (Experimental)
  Interventions: Drug: ALMB-0168

INTERVENTIONS:
Drug: ALMB-0168 — ALMB-0168 will be administered intravenously until either the disease progresses or intolerable toxicity occurs.

SUMMARY:
Bone metastasis is a common disease of advanced tumors. It refers to the metastasis of malignant tumors originating in a certain organ to the bones through the blood circulation or lymphatic system. The incidence of bone metastasis in breast and prostate cancer is as high as 65%-75%. Bone metastasis of malignant tumors often leads to severe bone lesions, including bone pain, pathological fractures, spinal cord compression, hypercalcemia and other bone-related events (SRE). SRE caused by bone metastasis of tumors can greatly reduce the quality of life of tumor patients. In severe cases, it can lead to rapid deterioration of the condition or even death, which greatly affects the extension of the patient's survival period. ALMB-0168 is designed to activate Cx43 hemichannels, which release key anti-cancer factors (such as ATP) into the extracellular environment. In several mouse models of breast cancer bone metastasis and orthotopic osteosarcoma, ALMB-0168 dose-dependently inhibited tumor growth and was able to extend the lifespan of tumor-bearing animals, indicating its potential as a therapeutic drug for malignant bone tumors. . Clinical research data from China and Australia show that ALMB-0168 is safe and initially effective in patients with bone metastasis and osteosarcoma;

DETAILED DESCRIPTION:
Avoid duplicating information that will be entered elsewhere, such as Eligibility Criteria or Outcome Measures.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically or cytologically pathologically confirmed solid tumors.
2. presence of any of the following:

   a. Cohort A breast cancer with bone metastases: patients with disease progression or intolerance to prior standard therapy (e.g., radiotherapy, chemotherapy, endocrine therapy, anti-Her2 targeted therapy) and the presence of bone metastatic lesions only.

   Among them, Cohort A needs to fulfill the following points:

   i. For hormone receptor-positive breast cancer: endocrine therapy (including, but not limited to, ET with or without combination of CDK 4/6 inhibitors, the mTOR inhibitor everolimus, the HDAC inhibitor cedarbenamide, and the PI3Kα inhibitor Alpelisib, among others) is required and progression or intolerance; ii. For Her2-positive (defined as FISH/CISH/SISH positive or IHC 3+ or IHC 2+ but confirmed HER2-positive by in situ hybridization) breast cancers: anti-Her2 targeted therapies (including trastuzumab/patuzumab or marketed biosimilars or initumumab or anti-Her2 ADCs such as T-DM1/DS8201 or TKIs) are required. DS8201 or TKI analogs (lapatinib, pyrrolitinib, neratinib, tucatinib, etc.)) and progression or intolerance; iii. For BRCA1/2 germline mutant breast cancer: progression or intolerance to olaparib is required; iv. PD-L1-positive with combined positive (CPS) score ≥10 requiring anti-PD-1, PD-L1 progression or intolerance; v. Disease progression or intolerance from at least 1 chemotherapy regimen, or unsuitable for chemotherapy; b. Cohort B prostate cancer with bone metastases: metastatic desmoplasia-resistant prostate cancer that meets PCWG3 progression criteria after prior standard therapy (e.g., docetaxel or abiraterone, enzalutamide, etc.), and the presence of bone metastatic lesions (≥2) only.

   Of these, Cohort B needs to fulfill the following points:

   i. Receiving or maintaining androgen deprivation therapy (ADT) during the study period (i.e., ongoing treatment with gonadotropin-releasing hormone (GnRH) agonists or antagonists (pharmacologic depot) or previous bilateral orchiectomy (surgical depot)), and serum testosterone must be at depot levels (< 50 ng/mL or < 1.7 nmol/L); ii. Must have progressed or been intolerant to at least 1 novel endocrine therapy (including enzalutamide/abiraterone/apatadine/darotarolimide, etc.) during the mCRPC phase; iii. Have received 1 paclitaxel-based chemotherapy regimen disease progression or intolerance, or are not suitable to receive paclitaxel.
3. 18 years old and above, male and female.
4. ECOG (Eastern Cooperative Oncology Group) PS score of 0, 1, or 2.
5. Major systemic functions are defined as follows:

   i. Bone marrow reserve: Absolute neutrophil count (ANC) ≥ 1.5 x 109/L; platelet count ≥ 75 x 109/L; hemoglobin ≥ 90 g/L, and no related supportive therapy such as GCS-F, EPO, or transfusion had been used in the 14 days prior to dosing; ii. Liver function: Total bilirubin ≤ 1.5 times the upper limit of normal (ULN) (unless the patient has grade 1 bilirubin elevation due to Gilbert's disease or a similar syndrome of slow bilirubin binding). Transaminases (AST/SGOT and/or ALT/SGPT) ≤ 3 times ULN; iii.Renal function: Normal serum creatinine ≤ 1.5 mg/dL (133 μmol / L) and calculated creatinine clearance ≥ 60 mL/min (Cockroft - Gault formula); iv. Coagulation: Coagulation parameters defined as an international normalized rate (INR) ≤ 2.

6 Eligible individuals of childbearing potential (males and females) must agree to use a reliable method of contraception (hormonal contraceptives, barrier method, or abstinence) with their partner for the duration of the trial and for at least 60 days after the last dose. Female individuals of childbearing age must have a negative blood pregnancy test within 7 days prior to enrollment and must be non-lactating. Male subjects are prohibited from donating sperm during their participation in the study and female subjects are prohibited from donating eggs during the study.

7. Expected survival of ≥ 3 months. 8. Be able to understand the whole process of the study, participate voluntarily and sign the informed consent form.

Exclusion Criteria:

1. Clinically uncontrolled pleural effusion, abdominal effusion, pericardial effusion (except for small amounts detected by imaging) within 4 weeks prior to dosing.
2. Poorly controlled bone pain, pathologic long bone fracture (> 50% cortical erosion on imaging), or neoplastic spinal cord compression.
3. Systemic glucocorticoid therapy within 4 weeks prior to dosing (except >20 mg/day of prednisone or equivalent dose of other hormones for prevention of contrast reactions during radiologic exams or inhalation or topical administration).
4. Following cardiac conditions within 6 months prior to dosing:

   1. Left ventricular ejection fraction (LVEF) < 45% as measured by echocardiography (ECHO);
   2. Screening electrocardiogram (ECG) suggesting a QTcF interval > 470 ms in women and > 450 ms in men;
   3. Unstable angina;
   4. Congestive heart failure (New York Heart Association [NYHA] > class 2);
   5. Acute myocardial infarction;
   6. Poorly controlled arrhythmias;
   7. Stent implantation.
5. Uncontrolled hypertension. (Systolic blood pressure > 160 mmHg or diastolic blood pressure > 100 mmHg.
6. Severe active bacterial, fungal, or viral infection (defined as requiring intravenous antibacterial, antifungal, or antiviral drug therapy) within 2 weeks prior to the first dose, or other serious medical condition that would interfere with the subject's ability to receive the test drug.
7. Positive anti-human immunodeficiency virus antibody or anti-syphilis spirochete-specific antibody tests, or active hepatitis B (defined as hepatitis B surface antigen positive and HBV-DNA above the lower measurable limit or ≥ 500 IU/ml) or active hepatitis C (defined as HCV antibody positive and HCV-RNA positive).
8. Other active tumors or a history of treatment for invasive tumors within 3 years. Subjects with a history of definitive local therapy for stage I tumors that are considered unlikely to recur are acceptable. Patients with a history of prior treatment for carcinoma in situ (e.g., non-invasive) and a history of non-melanoma skin cancer may be accepted.
9. Recent antineoplastic therapy (including but not limited to chemotherapy, immunotherapy, endocrine therapy and targeted therapy, but also including unlisted antineoplastic therapy) ≤ 4 weeks or within 5 half-lives of the drug, whichever is shorter, prior to the first dose, or relevant side effects NCI CTCAE v5.0 > Grade 1, except alopecia.
10. Participation in a clinical trial of another drug within 4 weeks prior to the first dose or within 5 half-lives of the trial drug, whichever is shorter, and enrollment in treatment, unless it is an observational (non-interventional) clinical trial or in the follow-up period of an interventional trial.
11. Radiation therapy (including radioisotope therapy such as strontium 89) ≤ 4 weeks prior to the first dose or localized radiation therapy ≤ 1 week prior to treatment, or have not recovered from the side effects of such therapy.
12. Surgery within 4 weeks prior to the first dose or outpatient surgery within 1 week prior to the start of treatment. There is no waiting period after artificial blood vessel placement.

13．Herbal or proprietary Chinese medicine with antitumor activity within 1 week prior to the first dose; 14. Previous grade ≥ 3 hypersensitivity and/or contraindications to human monoclonal antibodies or fusion proteins; 15. Pregnant or lactating women. 16. Individuals who, in the opinion of the investigator, are otherwise unsuitable for participation in this clinical trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 144 (Estimated)
Dates: Start 2024-05 (Estimated); Primary Completion 2026-06 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
The 6-month progression-free survival rate (6m-PFSR) of cohort A breast cancer IRC assessed according to RECIST 1.1 criteria | From date of randomization until the date of first documented progression or date of death from any cause, whichever came first, up to approximately 3 years
  time (in months) from enrollment to occurrence of any one of following: radiological tumor progressions using response evaluation criteria in solid tumors (RECIST 1.1), progression of bone lesions using Prostate Cancer Working Group 3 (PCWG2) criteria or occurrence of death due to any cause. Progression as per RECIST 1.1: at least a 20 percent (%) increase in sum of diameters of target lesions, unequivocal progression of existing non-target lesions. Progression of bone lesions (PCWG3 criteria): first bone scan with >= 2 new lesions compared to Baseline observed less than (<) 12 weeks from enrollment and confirmed by a second bone scan performed >=6 weeks; first bone scan with >=2 new lesions compared to Baseline observed >=12 weeks from enrollment
The 4-month progression-free survival rate (6m-PFSR) assessed by cohort B prostate cancer Independent Review Committee（IRC） based on PCWG 3 criteria Progression-free survival rate (4m-PFSR); | From date of randomization until the date of first documented progression or date of death from any cause, whichever came first, up to approximately 3 years
RP2D | From date of randomization until the date of first documented progression or date of death from any cause, whichever came first, up to approximately 3 years
  To determine the recommended Phase 2 dose (RP2D) of single agent ALMB-0168 (monotherapy) for further exploration

CONTACTS AND LOCATIONS:
Overall Officials: Jingnan Shen, M.D., Principal Investigator — First Affiliated Hospital, Sun Yat-Sen University

IPD SHARING:
Plan to Share IPD: No